CLINICAL TRIAL: NCT04476927
Title: Collecting and Evaluating Data of Potential Volatile Biomarkers in the Exhaled Air of Subjects With and Without COVID-19 by DiaNose
Brief Title: Detection of COVID-19 Subjects Using DiaNose Exhalation Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanose Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CORON01
Record Dates: First submitted 2020-06-16; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Total of 300 subjects - 200 suspected to COVID-19 and 100 healthy volunteers. all subjects will be undergo the DiaNose test.
  For data analysis and algorithm building, subjects will be divided into one of the following study groups:
  * Group 1: Covid-19 infected suspected (up to 300 subjects)
    * Sub-Group A: Clinical symptomatic patients with positive Covid-19 test (positive PCR);
    * Sub-Group B: Asymptomatic patients with positive Covid-19 test (positive PCR)
    * Sub-Group C: Clinical symptomatic patients with negative Covid-19 test (negative PCR) Additional sub-groups may be added according to clinical symptoms.
  * Group 2: Healthy volunteers (up to 100 subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- DiaNose procedure (Experimental): all subjects will be required to undergo the DiaNose exhalation test.
  Interventions: Device: DiaNose

INTERVENTIONS:
Device: DiaNose — DiaNose system is an electronic nose device that can "smell" diseases in the exhaled breath of patients in real time. The recognition of Volatile Organic Compounds (VOCs) in breath samples approach is non-invasive and for safe diagnosis of diseases.
  The DiaNose prototype system consists the following elements:
  * A Soft Tube connected to a Sensors Chamber - The soft tube is made of medical grade silicon. The subject blows air into the tube for a few seconds and the exhaled air is directed through the sensors chamber. This unit is for single use.
  * Sensors Reading Unit- a multi used unit for sensors signals measurement. The Sensor Reading Unit is connected to a Laptop either via a Data Acquisition Instrument - Commercial unit for resistance measurements (https://www.tek.com/keithley-switching-and-data-acquisition-systems/keithley-daq6510) (option A ) or directly by a USB cable (option B).
  * Laptop - Laptop is used to activate and save the test measurements.

SUMMARY:
The study aim is to collect and analyze data of potential Volatile Organic Compounds (VOCs) that could be used for discriminating between patients with and without COVID-19 or with high-risk for COVID-19 by DiaNose breath test.

up to 300 subjects will be enrolled to the study ( 200 COVID-19 suspected and 100 healthy volunteers in two clinical sites (1 in Israel and 1 in US).

DiaNose system is an electronic nose device that can "smell" diseases in the exhaled breath of patients in real time. This approach is non-invasive, simple and save.

The DiaNose prototype system consists the following elements:

A Soft Tube connected to a Sensors Chamber - The soft tube is made of medical grade silicon. The subject blows air into the tube for a few seconds and the exhaled air is directed through the sensors chamber. This unit is for single use.

• Sensors Reading Unit- a multi used unit for sensors signals measurement. The Sensor Reading Unit is connected to a Laptop that is used to activate and save the test measurements.

DETAILED DESCRIPTION:
This study is a prospective, multi-center research clinical study. The aim of this study is to collect and analyze data of potential Volatile Organic Compounds (VOCs) that could be used for discriminating between patients with and without COVID-19 or with high-risk for COVID-19 by DiaNose. The VOC profile of exhaled breath from subjects with COVID-19 infected suspected; and healthy volunteers, will be collected and analyzed to build and validate a predictive algorithmic model for diagnosing COVID 19.

Subjects which are COVID-19 infected suspected (Group 1); and healthy volunteers (Group 2), will be the study population. The study will encompass a total of up to 300 patients.

The COVID-19 infected suspected study group will be divided for the data analyzing and algorithm building into the following sub-groups (up to 200 subjects):

* Sub-Group A: Clinical symptomatic patients with positive Covid-19 test (positive PCR);
* Sub-Group B: Asymptomatic patients with positive Covid-19 test (positive PCR)
* Sub-Group C: Clinical symptomatic patients with negative Covid-19 test (negative PCR) Additional sub-groups may be added according to clinical symptoms. Up to 100 will be enrolled to the Healthy volunteers' study group. Subjects who meet general entry criteria will be asked to sign the study-specific Informed Consent Form the patient will be required not to eat/ smoke/ chewing gum or drink beverage other than water for one hour prior to the DiaNose exhalation test.

The patient will be asked to blow air into a disposable tube for a few seconds. Subject may be re-enrolled in case of need to perform additional PCR test and/or breath test with DiaNose according to standard of care or due to the study needs.

It is anticipated that it will require approximately 12 months to complete active enrollment.

ELIGIBILITY:
Inclusion Criteria:

Corona Suspected Subjects

1. Subject ≥18 years of age
2. Verified exposure to COVID-19 virus
3. Physical or Radiological evidence of Pneumonia or other Upper Respiratory Tract Infection
4. Subject with at least one of the following symptoms: Fever >37.80c P.O with no alternative source for infection / Cough / Nasal discharge or congestion / Shortness of breath (subjective or objective) with no alternative explanation / Sore throat / Loss of taste and smell / Combination of headache, general malaise, fatigue or other nonspecific URTI (upper respiratory tract infection) symptoms / GI symptoms (not as a signal symptom)
5. Subject has undergone PCR test or is about to undergo the test immediately
6. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
7. Subject is able and willing to adhere to the required testing

Exclusion Criteria:

1. Subject with HIV
2. Subject addicted to alcohol and/or drugs
3. Subject with active gingivitis
4. Subject with COPD (Chronic Obstructive Pulmonary Disease)
5. During the last hour before examination the subject ate including chewing gum / smoked/ Drank (any drink beside water)/performed excessive physical activity
6. Subject is pregnant (confirmed by subject declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
collecting and analyzing of DiaNose sensors signals from potential VOC markers in the breath samples of all subjects to build and validate a predictive algorithmic model for diagnosing COVID 19. | 1 hour
  Sensing Features (SFs) extracted from each of the sensors are used for statistical analysis by artificially intelligent/pattern recognition algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Peled, Study Director — Nanose Medical